CLINICAL TRIAL: NCT02659345
Title: Evaluating the Effectiveness of Art Therapy on Mood, Anxiety, and Pain Levels in Cancer Patients Undergoing Chemotherapy Treatment
Brief Title: Evaluating the Effectiveness of Art Therapy on Mood, Anxiety, and Pain Levels in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5Z15
Record Dates: First submitted 2016-01-14; First posted 2016-01-20 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Cancer
Keywords: Art Therapy; Chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Art Therapy (Experimental): The art therapy intervention will be executed by an art therapist at the Cancer Center. The same art therapy practices that are utilized in daily practice will be employed in this study. The intervention will include assessment of patient's needs and goals in addition to utilization of various art modalities. Sessions will conclude with processing of the art and supportive counseling as appropriate. Pilot testing of the intervention has been performed informally at Maroone Cancer Center with positive feedback provided by patients and their support systems to the physicians, nurses, and art therapist. Change in pain, emotional distress, depression, adn anxiety will be measured by the emotions thermometer.
  Interventions: Behavioral: Emotions Thermometer; Behavioral: Art Therapy

INTERVENTIONS:
Behavioral: Emotions Thermometer — The Emotions Thermometer, was chosen to assess patients' mood, anxiety level, and pain scale for this study. For patient ease, the study team chose to utilize a scale of 1-10 for all subjective measurements to be obtained from patients (mood and anxiety level). The study team included the thermometer image to mirror the NCCN Guidelines Version Distress Management Screening tool, for measuring distress and mood level. This screening tool has been shown to be effective in assessing patient distress and mood in oncology patients with ease of use in patients and utility in providers.
Behavioral: Art Therapy — Each participant will participate in a private art therapy session with the Art Therapist for 50 minutes. The participant will have a choice of materials to work with, including painting, drawing, clay, and collage materials. The session will conclude with processing of the art and supportive counseling.

SUMMARY:
Participants in this research study are asked to tell about their experience with art therapy. Participants in this research study are currently receiving chemotherapy treatment for cancer. The purpose of this study is to learn how art therapy affects mood, anxiety, pain, and emotions of individuals with cancer who are undergoing chemotherapy.

DETAILED DESCRIPTION:
In this single-center single-arm non-controlled descriptive study, we aim to describe the effects of a single art therapy session on a cancer patient's mood, pain, anxiety level.

Primary Objectives

* To assess the effect of art therapy on the cancer patient's mood
* To assess the effect of art therapy on the cancer patient's anxiety
* To assess the effect of art therapy on the cancer patient's pain

Secondary Objectives

* To explore differences in response to art therapy by ethnic group, race, age, sex, caregiver support, cancer diagnosis, reason for visit, and marital status
* To explore differences in response to art therapy by primary concern expressed by patients during art therapy sessions

ELIGIBILITY:
Inclusion Criteria:

* Subjects are able to give informed consent
* Any cancer diagnosis
* Actively undergoing any chemotherapy treatment at Maroone Cancer Center
* Patients who have never utilized art therapy at Maroone Cancer Center
* Speaks, reads, and writes in English
* Able and willing to participate in an art therapy session at Maroone Cancer Center

Exclusion Criteria:

* Patients without cancer diagnosis
* Patients not actively undergoing chemotherapy at Maroone Cancer Center
* Individuals unable to complete art therapy activities independently due to physical and/or mental impairment
* Under 18 years of age (minors)
* Patients who have dementia or a legal guardian
* Unable to speak, read, and write in English
* Patients who have previously utilized art therapy at Maroone Cancer Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01-25 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
The effect of art therapy on the cancer patient's mood | Change from baseline to after intervention, about 50 minutes
  The primary endpoint of the trial is to access the effect of an art therapy session on the patients' mood, anxiety level, and pain. To accomplish this, patients will complete four visual analog scales (VAS) prior to and after the session. The primary end points are the pre-and post session changes in the VAS.
The effect of art therapy on the cancer patient's anxiety | Change from baseline to after intervention, about 50 minutes
  The primary endpoint of the trial is to access the effect of an art therapy session on the patients' mood, anxiety level, and pain. To accomplish this, patients will complete four visual analog scales (VAS) prior to and after the session. The primary end points are the pre-and post session changes in the VAS.
The effect of art therapy on the cancer patient's pain | Change from baseline to after intervention, about 50 minutes
  The primary endpoint of the trial is to access the effect of an art therapy session on the patients' mood, anxiety level, and pain. To accomplish this, patients will complete four visual analog scales (VAS) prior to and after the session. The primary end points are the pre-and post session changes in the VAS.

SECONDARY OUTCOMES:
exploratory assessment of the association between sum of pain, anxiety, and mood visual analog scale (VAS) scores and ethnic group of patients | Change from baseline to after intervention, about 50 minutes
  The secondary goal is to assess, in an exploratory manner, associations between VAS scores (baseline and changes) and patient characteristics as well as patients' expressed primary concerns. Data will be analyzed using methods such as 2-sample and paired t-tests, ANOVA, and Pearson correlations.
exploratory assessment of the association between sum of pain, anxiety, and mood visual analog scale (VAS) scores and race of patients | Change from baseline to after intervention, about 50 minutes
  The secondary goal is to assess, in an exploratory manner, associations between VAS scores (baseline and changes) and patient characteristics as well as patients' expressed primary concerns. Data will be analyzed using methods such as 2-sample and paired t-tests, ANOVA, and Pearson correlations.
exploratory assessment of the association between sum of pain, anxiety, and mood visual analog scale (VAS) scores and age of patients | Change from baseline to after intervention, about 50 minutes
  The secondary goal is to assess, in an exploratory manner, associations between VAS scores (baseline and changes) and patient characteristics as well as patients' expressed primary concerns. Data will be analyzed using methods such as 2-sample and paired t-tests, ANOVA, and Pearson correlations.
exploratory assessment of the association between sum of pain, anxiety, and mood visual analog scale (VAS) scores and sex of patients | Change from baseline to after intervention, about 50 minutes
  The secondary goal is to assess, in an exploratory manner, associations between VAS scores (baseline and changes) and patient characteristics as well as patients' expressed primary concerns. Data will be analyzed using methods such as 2-sample and paired t-tests, ANOVA, and Pearson correlations.
exploratory assessment of the association between sum of pain, anxiety, and mood visual analog scale (VAS) scores and caregiver support of patients | Change from baseline to after intervention, about 50 minutes
  The secondary goal is to assess, in an exploratory manner, associations between VAS scores (baseline and changes) and patient characteristics as well as patients' expressed primary concerns. Data will be analyzed using methods such as 2-sample and paired t-tests, ANOVA, and Pearson correlations.
exploratory assessment of the association between sum of pain, anxiety, and mood visual analog scale (VAS) scores and cancer diagnosis of patients | Change from baseline to after intervention, about 50 minutes
  The secondary goal is to assess, in an exploratory manner, associations between VAS scores (baseline and changes) and patient characteristics as well as patients' expressed primary concerns. Data will be analyzed using methods such as 2-sample and paired t-tests, ANOVA, and Pearson correlations.
exploratory assessment of the association between sum of pain, anxiety, and mood visual analog scale (VAS) scores and reason for visit of patients | Change from baseline to after intervention, about 50 minutes
  The secondary goal is to assess, in an exploratory manner, associations between VAS scores (baseline and changes) and patient characteristics as well as patients' expressed primary concerns. Data will be analyzed using methods such as 2-sample and paired t-tests, ANOVA, and Pearson correlations.
exploratory assessment of the association between sum of pain, anxiety, and mood visual analog scale (VAS) scores and marital status of patients | Change from baseline to after intervention, about 50 minutes
  The secondary goal is to assess, in an exploratory manner, associations between VAS scores (baseline and changes) and patient characteristics as well as patients' expressed primary concerns. Data will be analyzed using methods such as 2-sample and paired t-tests, ANOVA, and Pearson correlations.
exploratory assessment of the association between sum of pain, anxiety, and mood visual analog scale (VAS) scores and primary concern expressed by patients during art therapy session | Change from baseline to after intervention, about 50 minutes
  The secondary goal is to assess, in an exploratory manner, associations between VAS scores (baseline and changes) and patient characteristics as well as patients' expressed primary concerns. Data will be analyzed using methods such as 2-sample and paired t-tests, ANOVA, and Pearson correlations.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Roshon, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Maroone Cancer Center - Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No